CLINICAL TRIAL: NCT05824234
Title: Multicenter Study on the Implementation of a Training Program in the Orientation of Care Towards Recovery (REFOCUS) in Mental Health Services
Brief Title: Implementation of REFOCUS Training Program in Mental Health Services
Acronym: RETAFORM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2021-A03025-36
Record Dates: First submitted 2023-03-28; First posted 2023-04-21 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, with cluster randomization with sequential permutation or stepped wedge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm number one (2023) (Other): Arm number one: services formed the first year with the REFOCUS formation Arm number two: services formed the second year with the REFOCUS formation Stepped wedge methodology
  Interventions: Other: Implementation of a training centered around the notions of recovery with mental health services first year
- Arm number two (2024) (Other): Arm number one: services formed the first year with the REFOCUS formation Arm number two: services formed the second year with the REFOCUS formation Stepped wedge methodology
  Interventions: Other: Implementation of a training centered around the notions of recovery with mental health services second year

INTERVENTIONS:
Other: Implementation of a training centered around the notions of recovery with mental health services first year — Stepped wedge design so same procedure for both arms Stepped-wedge design with randomization stratified by cluster (training over the 1st or 2nd year) according to professional practice (intra-hospital, CMP / CATTP, day hospital, Psychosocial Rehabilitation Center, mobile team, medical sector) social) of the teams formed by the 18 centers participating in the study
  Arms: Arm number one (2023)
Other: Implementation of a training centered around the notions of recovery with mental health services second year — Stepped wedge design so same procedure for both arms Stepped-wedge design with randomization stratified by cluster (training over the 1st or 2nd year) according to professional practice (intra-hospital, CMP / CATTP, day hospital, Psychosocial Rehabilitation Center, mobile team, medical sector) social) of the teams formed by the 18 centers participating in the study
  Arms: Arm number two (2024)

SUMMARY:
Training of mental health service teams in the orientation of care towards recovery through a 3-day training course: REFOCUS. This training aims to orient care towards recovery. Following this training, evaluation of the effectiveness of the implementation of REFOCUS training in mental health services.

DETAILED DESCRIPTION:
The primary hypothesis is that the implementation of REFOCUS will facilitate the 1-year recovery of patients managed by trained professionals. The secondary hypotheses are that the implementation of REFOCUS will facilitate improved orientation of practices towards recovery; reduced costs associated with the use of mental health services; improved perceived stigma, self-stigma, stigma-related stress, well-being, perceived coercion, and general functioning among those involved.

ELIGIBILITY:
Inclusion Criteria:

* Age from 15 to 65 years old.
* Diagnosis of schizophrenia, schizoaffective disorder, schizotypal disorder and schizophreniform disorder or bipolar disorder, borderline personality disorder, disabling anxiety or depressive disorder (DSM-V criteria; APA, 2013).
* Patients cared for by the team or unit benefiting from REFOCUS training
* French mother tongue.
* Patient affiliated or entitled to a social security scheme
* Patient having received information about the study and having confirmed their participation in the study by signing the consent form
* For minors (< 18 years), information given to holders of parental authority and signature of consent.
* For patients under curatorship, form signed by the patient and information given to the curator

Exclusion Criteria:

* Age less than 15 years old
* Patients under guardianship
* Presence of an associated intellectual disability
* Neurological disorders of vascular, infectious or neurodegenerative origin.
* Taking somatic drugs with a cerebral or psychic impact (eg corticosteroids).

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire about the Process of Recovery QPR Intra- and inter-group comparison in users with severe psychiatric disorders | Two years
  Intra- and inter-group comparison of the score on the self-assessment scale of the stage of recovery (Questionnaire about the Process of Recovery; QPR) in users with severe psychiatric disorders The QPR has 15 items each scored on a 4-point scale (0= disagree strongly, 1=disagree, 2=neither agree nor disagree, 3=agree, 4=agree strongly). Higher scores are indicative of recovery. However, those involved in developing this measure suggest that scores should not only be added to give total scores, but the QPR should be used as described above e.g. as a tool for considering personal goals for recovery, health and wellbeing.

SECONDARY OUTCOMES:
Recovery Self-Assessment (RSA) health professional version to assess the perception of having a recovery-oriented practice | One year
  Intra- and inter-group comparison of scores on the following scales:
  The Recovery Self-Assessment (RSA) is a 36-item measure designed to gauge the degree to which programs implement recovery-oriented practices. It is a self-reflective tool designed to identify strengths and target areas of improvement as agencies and systems strive to offer recovery-oriented care.
Self-stigma scale (Internalized Stigma of Mental Illness) | One year
  Intra- and inter-group comparison of scores on the following scale
Warwick-Edinburgh Mental Well Being Scale (WEMWBS) for mental well-being | One year
  Intra- and inter-group comparison of scores on the following scale Scoring. The 14-item scale WEMWBS is very simple to score. The total score is obtained by summing the score for each of the 14 items. The scoring range for each item is from 1 - 5 and the total score is from 14-70.
Qualitative component | Two years
  A qualitative analysis will be conducted with trainers, trained mental health professionals and patients followed by trained professionals, using semi-structured individual interviews or focus groups. For this study, participants will be asked about their experience following the implementation of REFOCUS training in recovery-oriented practices. The focus groups will be facilitated by at least two members of the research team, recorded with the participants' consent and fully transcribed. They will be conducted until data saturation is achieved. The data will be analysed using the thematic content analysis method. The COREQ grid will be used to write the protocol and analyse the results. Multiple triangulation of the data will help to refine the understanding of the problem and limit the risk of interpretation bias

CONTACTS AND LOCATIONS:
Overall Officials: Julien DUBREUCQ, PH, Principal Investigator — CHU ST ETIENNE
Locations (1):
- centre de réhabilitation - Hôpital le Vinatier, Lyon, Rhône, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dubreucq J, Franck N, Plasse J, Muller AE, Bralet MC, Bera-Potelle C, Berna F, Blachere C, Carpentier A, Chereau I, Chillet P, Dubreucq M, Durand-Zaleski I, Chirio-Espitalier M, Espi P, Fourneret P, Gabriel-Segard T, Guioux A, Grange AL, Green A, Green E, Guillard-Bouhet N, Gerardin P, Harscoet YA, Khazaal Y, Lassere E, Le Bras A, Leamy M, Legrand G, Legros-Lafarge E, Llorca PM, Jaafari N, Mabille L, Masson D, Massoubre C, Moisset A, Nahabedian N, Quiles C, Reydellet D, Simon A, Sibert A, Tresse R, Tinland A, Meadows G, Slade M; RETAFORM study group. Evaluation of a pro-recovery training intervention (REFOCUS-RETAFORM) in specialist mental health services across France: stepped-wedge cluster randomised controlled trial protocol. BMC Psychiatry. 2025 Oct 14;25(1):982. doi: 10.1186/s12888-025-07253-w. PMID 41088104